CLINICAL TRIAL: NCT01322139
Title: A Multiple-Dose, Randomized, Double-Blind, Placebo- and Active-Controlled, Four-Arm, Parallel Group Thorough QT/QTc Study to Evaluate the Electrophysiologic Effects of Sativex.
Brief Title: Sativex Thorough QT/QTc Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GWCP0607
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Effects of Sativex on ECG
Keywords: Sativex; Cannabinoid; Electrocardiogram; QT interval
MeSH Terms: conditions — Marijuana Abuse | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High dose placebo and oral moxifloxacin placebo (Placebo Comparator): 24 or 36 placebo sprays (12 or 18 sprays twice daily) for 5 days and single oral moxifloxacin placebo on Day 5.
  Interventions: Drug: Placebo spray and oral moxifloxacin placebo
- Low dose Sativex and oral moxifloxacin placebo (Active Comparator): 8 Sativex sprays (4 sprays twice daily) + 16 or 28 placebo sprays (8 or 14 sprays twice daily) for 5 days and single oral moxifloxacin placebo on Day 5.
  Interventions: Drug: Sativex spray and oral moxifloxacin placebo
- High dose Sativex and oral moxifloxacin placebo (Active Comparator): 24 or 36 Sativex sprays (12 or 18 sprays twice daily) for 5 days and single oral moxifloxacin placebo on Day 5.
  Interventions: Drug: Sativex spray and oral moxifloxacin placebo
- High dose placebo and single oral moxifloxacin 400 mg tablet (Active Comparator): 24 or 36 placebo sprays (12 or 18 sprays twice daily) for 5 days and single oral moxifloxacin 400 mg tablet on Day 5.
  Interventions: Drug: Placebo spray and moxifloxacin

INTERVENTIONS:
Drug: Placebo spray and oral moxifloxacin placebo — 24 or 36 placebo sprays (12 or 18 sprays twice daily every 12 hours) for 5 days and single oral moxifloxacin placebo on Day 5.
  Arms: High dose placebo and oral moxifloxacin placebo
Drug: Sativex spray and oral moxifloxacin placebo — 8 Sativex sprays (4 sprays twice daily every 12 hours) + 16 or 28 placebo sprays (8 or 14 sprays twice daily every 12 hours) for 5 days and single oral moxifloxacin placebo on Day 5.
  Arms: Low dose Sativex and oral moxifloxacin placebo
Drug: Sativex spray and oral moxifloxacin placebo — 24 or 36 Sativex sprays (12 or 18 sprays twice daily every 12 hours) for 5 days and single oral moxifloxacin placebo on Day 5.
  Arms: High dose Sativex and oral moxifloxacin placebo
Drug: Placebo spray and moxifloxacin — 24 or 36 placebo sprays (12 or 18 sprays twice daily every 12 hours) for 5 days and single oral moxifloxacin 400 mg tablet on Day 5.
  Arms: High dose placebo and single oral moxifloxacin 400 mg tablet

SUMMARY:
This study was to evaluate effects of Sativex on electrocardiogram (ECG) traces when administered at its therapeutic dose of 8 sprays per day and at multiples of the therapeutic dose (24 or 36 sprays per day), and to evaluate its safety and tolerability.

DETAILED DESCRIPTION:
This is a multiple-dose, randomized, double-blind, double-dummy, placebo- and active-controlled, four arm, parallel group study to evaluate the effect of Sativex on the QT/QTc interval.

Within 30 days of screening, eligible subjects were randomized to one of four treatment groups. Baseline ECG measurements were recorded at specified times and the following day, subjects commenced five days treatment with Sativex or placebo. On Day 5, subjects then received either moxifloxacin 400 mg (Group 4) or moxifloxacin placebo (Groups 1, 2 and 3). Triplicate ECG measurements and pharmacokinetic samples were collected on Day 5. On days 1-5, Safety ECG measurements were also collected at pre-dose and 2 hours post-dose. Subjects returned to the study centre for an outpatient safety follow-up visit approximately 10-14 days after their last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 18 to 45 years of age.
* Body Mass Index (BMI) within the range of 19 to 29.9 kg/m2, and a minimum weight of at least 50 kg at screening.
* Non-users of tobacco products (minimum of 6 months)
* Free from any clinically significant abnormality on the basis of medical history, vital signs, physical examination, ECG, and laboratory evaluation at screening and admission to the treatment session, as judged by the investigator or designee.
* Systolic blood pressure between 90 to 140 mmHg and diastolic blood pressure between 50 and 90 mmHg at screening and admission to the treatment session.
* Subjects with reproductive potential required to practice abstinence or be using and willing to continue using a medically acceptable form of birth control for at least one month prior to screening (at least 3 months for oral contraceptives) and for at least 60 days after the last study drug administration.
* Female subjects required to have a negative serum pregnancy test at screening and admission to the treatment session.
* Subjects must have been able to speak, read and understand English sufficiently to understand the nature of the study, to provide written informed consent, and to allow completion of all study assessments.
* Subjects must have understood and provided written informed consent prior to initiation of any protocol-specific procedures.
* Subjects must have been willing and able to abide by all study requirements and restrictions.

Exclusion Criteria:

* History or presence of drug or alcohol abuse or dependence (as determined by the Diagnostic and Statistical manual, 4th Revision [DSM-IV] for abuse and dependence), including subjects who had ever been in a drug rehabilitation program.
* Clinically significant abnormalities on oral or physical examination, medical history, ECG, vital signs, or laboratory values at screening or admission to the treatment session, as judged by the investigator or designee.
* Any known or suspected history (including family history) of schizophrenia or other psychotic illness. Presence or history of an organic brain disorder or seizure disorder deemed clinically significant by the investigator.
* History or presence of clinically significant pulmonary, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition, which in the opinion of the investigator would have jeopardised the safety of the subject or the validity of the study results.
* Known cardiovascular condition or history of a cardiovascular condition at screening.
* Pulse rate at rest less than 45 or greater than 100 beats per minute.
* Abnormal screening ECG indicating a second- or third-degree atrioventricular block, or one or more of the following: QRS greater than 109 msec, QTc greater than 450 msec, PR interval greater than 200 msec. Any rhythm other than sinus rhythm, which was interpreted by the investigator to be clinically significant.
* History of torsade de pointes or risk factors for torsade de pointes (e.g. heart failure, hypokalemia, family history of Long QT syndrome).
* Postural drop of 20 mmHg or more in systolic blood pressure at screening.
* Use of non-prescription drug within 7 days prior to the first drug administration (in particular iron and antacids). Subjects who had taken over-the-counter medication could still be entered into the study, if in the opinion of the investigator or designee, the medication received would not interfere with the study procedures or data integrity or compromise the safety of the subject.
* Use of any prescription medications (except acceptable forms of birth control and hormone replacement), natural health products, or recreational drugs within 14 days or 5 elimination half-lives (whichever was longer) prior to first drug administration or throughout the study, unless in the opinion of the investigator or designee, the product would not interfere with the study procedures or data integrity or compromise the safety of the subject. In particular medications that prolong the QT/QTc interval (e.g. erythromycin, antipsychotics, tricyclic antidepressants)were strictly avoided.
* Currently using cannabis or tetrahydrocannabinol (THC)-containing medicines (as shown by positive urine drug screen). Subjects who had used natural or synthetic cannabinoid based medications (including Sativex, Marinol or Acomplia [rimonabant]) within 3 months prior to study entry and were unwilling to abstain for the duration of the study.
* Habituation to analgesic drugs (i.e. routine use of oral analgesics 5 or more times per week).
* Positive urine drug screen upon presentation for screening or at admission to the treatment session.
* Positive breath alcohol test at screening or at admission to the treatment session.
* Female subjects who were pregnant or lactating or who were planning to become pregnant within 60 days of last study drug administration.
* Inability to refrain from consuming caffeine (including caffeine pills, cola, tea, coffee, energy drinks, or any other caffeinated product) for at least nine days.
* History of allergy or hypersensitivity to cannabinoids, propylene glycol, ethanol, peppermint oil, moxifloxacin or other quinolone antimicrobials, related drugs, or any of the drug excipients or other drug product components.
* Positive for Hepatitis B, Hepatitis C, or HIV at screening.
* Donation of 50 mL to 499 mL whole blood within 30 days or donation of more than 499 mL whole blood within 56 days of admission to the treatment session.
* Current or pending legal charges or currently on probation.
* Treatment with any investigational drug within 30 days prior to screening.
* Study site or Sponsor employee or relative of an employee who was directly involved in the study.
* A subject who, in the opinion of the investigator or designee, was not considered to be suitable and was unlikely to comply with the study protocol for any reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Time-matched change from baseline in QTc based on an individual correction (QTcl) | 5 days

SECONDARY OUTCOMES:
QTc with Fridericia correction method (QTcF) and the QTc with Bazett correction (QTcB) | 5 days
Heart Rate | 5 days
PR interval | 5 days
QRS interval | 5 days
Uncorrected QT interval | 5 days
Change in ECG morphological patterns | 5 days
Correlation between the QTcl change from baseline and plasma concentrations of the parent metabolites | 5 days
Adverse Events | Up to 2 weeks after final dose
Clinical laboratory parameters | Up to 2 weeeks after final dose
Vital signs | Up to 2 weeks after final dose
Oral and physical examination | Up to 2 weeks after final dose
Peak plasma concentration (Cmax) | Days 5 and 6
Time to peak plasma concentration (Tmax) | Days 5 and 6
Area under the concentration curve (AUC(0-t) and AUC(0-inf)) | Days 5 and 6

CONTACTS AND LOCATIONS:
Locations (1):
- DecisionLine Clinical Research Corporation, Toronto, Ontario, Canada

REFERENCES:
- [Result] Sellers EM, Schoedel K, Bartlett C, Romach M, Russo EB, Stott CG, Wright S, White L, Duncombe P, Chen CF. A Multiple-Dose, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group QT/QTc Study to Evaluate the Electrophysiologic Effects of THC/CBD Spray. Clin Pharmacol Drug Dev. 2013 Jul;2(3):285-94. doi: 10.1002/cpdd.36. Epub 2013 May 14. PMID 27121791